CLINICAL TRIAL: NCT04987450
Title: Effect of High-dose Glucocorticoids on Markers of Inflammation and Bone Metabolism in Patients With Primary Glomerular Disease
Brief Title: Effect of Glucocorticoids on Inflammation and Bone Metabolism in Patients With Glomerular Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Lodz (Other)
Responsible Party: Principal Investigator, Michal Nowicki, Professor, Medical University of Lodz
Other Study IDs: RNN/267/17/KE
Record Dates: First submitted 2021-07-22; First posted 2021-08-03 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-08

CONDITIONS: Glomerular Disease
Keywords: glucocorticoids; primary glomerular disease; sirtuin-1; sclerostin
MeSH Terms: conditions — Sclerosteosis | interventions — Methylprednisolone; Prednisone

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study population: Plasma levels of SIRT-1, IL-6, FGF-23, sclerostin, calcium, phosphate, PTH and urine excretion of total protein, albumin, creatinine, calcium and phosphate are measured at baseline. Then the patients receive three intravenous daily pulses of methylprednisolone of 500 mg followed by oral prednisone 0.8-1.0 mg/kg/24h. The same measurements are repeated 4, 7 and 30 days after starting the steroid treatment.
  Interventions: Drug: Methylprednisolone, prednisone

INTERVENTIONS:
Drug: Methylprednisolone, prednisone — The patients receive intravenous pulses of methylprednisolone 20-30 mg/kg/day for three consecutive days followed by oral prednisone 0.8-1.0 mg/kg/day.

SUMMARY:
The aim of the study is to assess the influence of high doses of intravenous corticosteroids on plasma inflammation and bone markers in patients with primary glomerular disease. The study would include 40 patients with chronic kidney disease. The main inclusion criterion is clinical and histopathological diagnosis of primary glomerular disease and urine protein excretion >2.0 g/24h. The exclusion criteria include secondary glomerular disease, acute kidney injury, acute or chronic inflammation, history of non-compliance.

DETAILED DESCRIPTION:
Glucocorticoids are one of the most widely used classes of drugs to treat inflammatory and autoimmune diseases. They increase formation of osteoclasts and enhance bone resorption thereby increasing risk of bone fractures and osteoporosis.

Sirtuin-1(SIRT-1) belongs to family of proteins involved in protection against inflammation and oxidative stress. A role of SIRT-1 in regulation of bone metabolism during high-dose steroid therapy is unknown.

The study protocol was approved by the local Bioethics Committee and the study is conducted according to the Declaration of Helsinki. Adult patients with the previous diagnosed primary glomerular disease based on both clinical and renal biopsy findings are included.

Plasma concentration of SIRT-1, interleukin-6 (IL-6), fibroblast growth factor 23 (FGF-23), sclerostin, calcium, phosphate, parathormone (PTH) and urine excretion of total protein, albumin, creatinine, calcium and phosphate are measured at baseline. Then the patients receive three intravenous pulses of methylprednisolone of 500 mg followed by oral prednisone 0.8-1.0 mg/kg/24h. The same measurements are repeated 4, 7 and 30 days after starting the steroid treatment.

ELIGIBILITY:
Inclusion Criteria:

* previous diagnosed primary glomerular disease based on both clinical and renal biopsy findings
* an estimated glomerular filtration rate ≥15 ml/min/1.73m2
* proteinuria ≥2.0 g/24h

Exclusion Criteria:

* secondary glomerular disease
* acute kidney injury
* acute or chronic inflammation
* malignancy
* uncontrolled hypertension with systolic blood pressure higher than 160 mmHg
* symptomatic hypotension
* advanced heart failure
* history of non-compliance, dementia or depression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients with primary glomerular disease who are diagnosed and hospitalized in Nephrology Department in Łódź.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2021-07-30 (Estimated); Study Completion 2021-07-30 (Estimated)

PRIMARY OUTCOMES:
the change of plasma SIRT-1 level after glucocorticoids administration | 30 days
the change of plasma sclerostin level after glucocorticoids administration | 30 days
the change of plasma FGF-23 level after glucocorticoids administration | 30 days
the change of plasma IL-6 level after glucocorticoids administration | 30 days
the change of plasma total calcium level after glucocorticoids administration | 30 days
the change of plasma phosphate level after glucocorticoids administration | 30 days
the change of plasma PTH level after glucocorticoids administration | 30 days
the change of urine albumin/creatinine ratio after glucocorticoids administration | 30 days
the change of urine total protein/creatinine ratio after glucocorticoids administration | 30 days
the change of urine phosphate/creatinine ratio after glucocorticoids administration | 30 days
the change of urine calcium/creatinine ratio after glucocorticoids administration | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Michał Nowicki, Prof. MD., Principal Investigator — Department of Nephrology, Hypertension and Kidney Transplantation Medical University of Lodz, Poland
Locations (1):
- Medical University of Lodz, Poland, Lodz, Poland

IPD SHARING:
Plan to Share IPD: No